CLINICAL TRIAL: NCT01344772
Title: Total Hip Arthroplasty Compared to Internal Fixation for Displaced Intracapsular Fractures of the Femoral Neck. A Randomized, Controlled Trial With a Seventeen Year Follow-up
Brief Title: Total Hip Arthroplasty Compared to Internal Fixation for Displaced Intracapsular Fractures of the Femoral Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Olof Skoldenberg, Consulatant Orthopaedic Surgeon, PhD, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19902010
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Femoral Neck Fracture
Keywords: femoral neck fracture; total hip arthroplasty; internal fixation
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Fracture Fixation, Internal; Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internal fixation (Active Comparator): Displaced femoral neck fracture treated with internal fixation using two parallel cannulated screws.
  Interventions: Procedure: Internal fixation
- Total hip replacement (Active Comparator): Displaced femoral neck fracture treated with total hip replacement through a posterior approach.
  Interventions: Procedure: Total hip arthroplasty

INTERVENTIONS:
Procedure: Internal fixation — Two cannulated screws are placed under x-ray guidance
  Arms: Internal fixation
Procedure: Total hip arthroplasty — A total hip arthroplasty is performed through a standard posterior approach
  Arms: Total hip replacement

SUMMARY:
The primary aim of this study was to determine the Harris hip score as an evaluation of hip function, in mentally competent elderly patients (>65 years old) treated with either THR or IF, after contracting a displaced femoral neck fracture. The secondary aim was to compare the rate of reoperations and complications between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Acute displaced femoral neck fracture Garden III or IV,
* Age over 65 years,
* Admission from their own home,
* No concurrent joint disease or previous fracture in the lower extremities,
* Healthy or controlled medical conditions without significant systemic effects (ASA 1-2),
* Harris hip score of 100
* Acceptance from the patient to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 1990-02; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Harris hip score | 17 years
  HHS index score of 0 indicates the worst possible function of the hip and a value of 100 indicates full function.

SECONDARY OUTCOMES:
Reoperations and complications | 17 years
  IF group: nonunion, osteonecrosis, deep infection or fracture in the vicinity of the screws. Protruding screws or extraction of the screws when the fracture was healed was not defined as a complication.
  THR group: radiographic signs of loosening of the femoral- or acetabular component, dislocation, periprosthetic fracture or deep infection

CONTACTS AND LOCATIONS:
Overall Officials: Olof Sköldenberg, MD, PhD, Principal Investigator — Danderyd Hospital
Locations (1):
- Danderyd Hospital, Stockholm, Sweden